CLINICAL TRIAL: NCT03503071
Title: Recovery of Quality of Life After Cytoreductive Surgery and Intraperitoneal Chemotherapy for Colorectal Cancer and Pseudomyxoma Peritonei
Brief Title: Quality of Life After Cytoreductive Surgery and Intraperitoneal Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Soo Yeun Park, Principal investigator, Kyungpook National University Hospital
Other Study IDs: KNUHC03
Record Dates: First submitted 2018-04-09; First posted 2018-04-19 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Cytoreduction Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cytoreductive surgery and intraperitoneal chemotherapy — Cytoreductive surgery and intraperitoneal chemotherapy for colorectal cancer or pseudomyxoma peritonei. Either early postoperative intraperitoneal chemotherapy (EPIC) or hyperthermic intraperitoneal chemotherapy (HIPEC) is used for intraperitoneal chemotherapy.

SUMMARY:
Cytoreductive surgery with intraperitoneal chemotherapy is one of the most important treatments for patients with colorectal cancer and peritoneal metastasis. For the best survival rates, complete removal of all metastatic lesions is the most important part of treatment, and various surgical procedures are required for the complete cytoreduction. Therefore, the postoperative morbidity rates are higher than those of localized colon cancer surgeries and patients can experience a prolonged recovery period and deterioration of physical activities over a long period. The aim of this study is to investigate the change of quality of life after cytoreductive surgery and intraperitoneal chemotherapy for colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer peritoneal metastasis
* Pseudomyxoma peritonei
* ECOG (Eastern Cooperative Oncology Group) performance status 0-3
* Normal bone marrow, kidney, and liver function
* Patient must sign and date the informed consent

Exclusion Criteria:

* Palliative surgery
* Palliative intraperitoneal chemotherapy
* Psychotic disorder
* Drug abuser

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for cytoreductive surgery and intraperitoneal chemotherapy for colorectal cancer peritoneal metastasis or pseudomyxoma peritonei
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Brief pain inventory (BPI) | Changes from baseline pain scores at postoperative 12 months
  Pain recovery after cytoreductive surgery and intraperitoneal chemotherapy

SECONDARY OUTCOMES:
European Organisation for Research and Treatment of Cancer (EORTC) Quality of life questionnaire (QLQ)-C30 | preoperative, postoperative 3 months, postoperative 6 months, postoperative 12 months, postoperative 24 months
  Qualify of life questionnaire for cancer patients
EORTC QLQ for colorectal cancer | preoperative, postoperative 3 months, postoperative 6 months, postoperative 12 months, postoperative 24 months
  Quality of life questionnaire for patients with colorectal cancer
Short-form(SF)-36 | preoperative, postoperative 3 months, postoperative 6 months, postoperative 12 months, postoperative 24 months
  Global measure of health-related quality of life
Postoperative morbidity | 90 days after surgery
  Incidence and degree of surgical and medical complications after surgery
Postoperative mortality | 90 days after surgery
  Incidence of postoperative mortality
Postoperative recovery | 150 days after surgery
  Duration of hospital stay after surgery
Brief pain inventory (BPI) | preoperative, postoperative 3 months, postoperative 6 months, postoperative 24 months
  Pain recovery after cytoreductive surgery and intraperitoneal chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Soo Yeun Park, MD, Principal Investigator — Colorectal Cancer Center, Kyungpook National University Chilgok Hospital
Locations (1):
- Kyungpook National University Chilgok Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No